CLINICAL TRIAL: NCT03872687
Title: An Evaluation of the Effectiveness of Single Tufted Brush in the Management of Peri-implant Mucositis in Healthy Individuals: A Randomised Controlled Single Blinded Clinical Trial
Brief Title: The Effectiveness of Single Tufted Brush in the Management of Peri-implant Mucositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Jia Hui Fu, Assistant Professor, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/01174
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Dental Implant
Keywords: dental implants, tufted brush, IDB, mucositis, gingivitis
MeSH Terms: conditions — Mucositis; Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single tufted brush with IDB (Experimental): Subjects in this group will receive a single tufted brush and interdental brushes of an appropriate size for 6 months.
  Interventions: Device: single tufted brush with IDB
- interdental brushes (Active Comparator): Subjects in this group will only receive interdental brushes 6 months.
  Interventions: Device: interdental brushes

INTERVENTIONS:
Device: single tufted brush with IDB — Subjects in this group will receive a single tufted brush and interdental brushes of an appropriate size that will fit the interdental spaces around the implant.
  Arms: single tufted brush with IDB
Device: interdental brushes — Subjects in this group will only receive interdental brushes
  Arms: interdental brushes

SUMMARY:
The study aims to investigate and compare the reduction in (1) soft tissue inflammation and (2) amount of plaque accumulation at implant sites with (test) or without (control) patient administered use of single tufted brush.

Stratified randomized single blinded clinical controlled trial with 2 parallel arms is designed to achieve the aims of this research project. Study participants will be enrolled from NUH University Dental Cluster. They will be randomly assigned into the test (toothbrush, interdental brush, and single tufted brush) and control (toothbrush and interdental brush) groups and reviewed at 2 weeks (± 3 days), 4 weeks (± 3 days), 3 months (± 7 days), and 6 months (± 7 days).

DETAILED DESCRIPTION:
There are two study phases during the whole course of the study. PHASE 1: EXAMINER CALIBRATION Examiner will be calibrated before the study period with 10 volunteers.

The intra-examiner reliability will be assessed using intraclass correlation coefficient. The volunteers will be recruited based on the inclusion and exclusion criteria.

Clinical Parameters:

i. Probing pocket depths (PPD) at 6 sites per implant ii. mBI at 6 sites per implant iii. mPI at 8 sites per implant Clinical parameters (i) to (iii) will be performed at day 0 and day 7.

PHASE 2: STUDY INTERVENTION Study participants who are visiting University Dental Cluster or any other dental clinics or hospitals will be referred for this study. They will be enrolled at NUH University Dental Cluster if they fulfill the inclusion and exclusion criteria.

Groups:

* Test: Subjects in this group will receive a single tufted brush and interdental brushes of an appropriate size that will fit the interdental spaces around the implant.
* Control: Subjects in this group will only receive interdental brushes.

Randomization:

Study subjects will be randomly assigned into either test or control group based on a computer generated randomization code after screening of inclusion and exclusion criteria and signing of informed consent form.

Blinding and Allocation Concealment:

The study examiner who will be doing the clinical examination and collecting the study data will be blinded to the group allocation; however it is not possible to blind the study subjects to the group allocation. The clinician, who will be performing the treatment and providing oral hygiene instructions, will be given a sequentially numbered envelope containing the subject's group allocation after non-surgical periodontal therapy has been performed and before giving the oral hygiene instructions.

Clinical Parameters:

i. Probing pocket depths (PPD) (6 points per implant) ii. mBI (6 points per implant) iii. mPI (8 points per implant) iv. Characteristics of the implant and implant crown: tissue level or bone level, supraor submucosal margin, degree of overcontour as seen on periapical radiograph v. Peri-apical radiograph of implant taken with parallel technique Clinical parameters (i) to (iii) will be performed at baseline, 2-weeks, 1 month, 3 months, and 6 months post instrumentation.

Clinical parameter (iv) and (v) will be performed at baseline.

Radiographic Analysis:

Peri-apical radiographs will be taken with paralleling technique to determine that there is peri-implant bone loss beyond 2mm at baseline.

ELIGIBILITY:
Inclusion Criteria:

i. Age 21-70 years old ii. Medically healthy (ASA I or II) iii. Presence of interdental spaces that will allow an interdental brush to pass through without soft tissue trauma iv. Single moderately rough tissue level or bone level dental implants, which were restored with single screw or cement retained crowns and in function for the past 2-5 years v. Implants should have peri-implant mucositis that is defined as (Renvert, et al., 2018)

* Presence of clinical signs of inflammation, which are redness, shininess of the soft tissue surface, local swelling, with or without increase in probing depth
* Bleeding on probing
* No progressive peri-implant bone loss beyond 2mm from implant platform (Rosen, et al., 2013) vi. Implants with at least 1mm of keratinized peri-implant mucosa

Exclusion Criteria:

i. Embrasure space between the implant and adjacent tooth is non-existent or too small to permit the use of an interdental brush ii. Self declared pregnancy iii. Heavy smokers (1 pack a day) iv. Uncontrolled or poorly controlled medical conditions e.g. diabetes (HBA1c 8.5% and above) v. Untreated oral conditions e.g. active periodontitis vi. On medications that will cause gingival enlargement vii. Any hyperplastic interdental papilla that will hinder interdental cleaning viii. Antibiotics intake within the past 3 months ix. Parkinson's disease and other debilitating diseases x. Subjects who are unable to give consent e.g. mentally challenged

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-06-07 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
the reduction in bleeding tendency | baseline, 2-weeks, 1 month, 3 months, and 6 months post instrumentation
  The reduction in bleeding tendency as assessed by mBI at 6 sites per implant

SECONDARY OUTCOMES:
the reduction in plaque accumulation | baseline, 2-weeks, 1 month, 3 months, and 6 months post instrumentation
  The reduction in plaque accumulation with a modified Plaque Index (mPI) at 8 sites (mesiobuccal, mesial, mesiolingual, lingual, distolingual, distal, distobuccal, and buccal) per implant

CONTACTS AND LOCATIONS:
Overall Officials: Jia Hui Fu, Master, Principal Investigator — National University Health System, Singapore

IPD SHARING:
Plan to Share IPD: No